CLINICAL TRIAL: NCT01154335
Title: A Phase I Study of Everolimus (mTOR Inhibitor) and OSI-906 (Dual IGFR and IR Tyrosine Kinase Inhibitor) for the Treatment of Patients With Refractory Metastatic Colorectal Cancer
Brief Title: Everolimus and OSI-906 for Patients With Refractory Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis Pharmaceuticals (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 124
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Results first posted 2015-01-14 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: refractory metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose Level 1 (Experimental): combination of OSI-906 and everolimus
  OSI-906: 50 mg Twice a Day, cycle-28 days
  Everolimus: 5mg Daily, cycle-28 days
  Interventions: Drug: OSI-906; Drug: Everolimus
- Dose Level 2 (Experimental): combination of OSI-906 and everolimus
  OSI-906: 100 mg Twice a Day, cycle-28 days
  Everolimus: 10mg Daily, cycle-28 days
  Interventions: Drug: OSI-906; Drug: Everolimus
- Dose Level 2a (Experimental): combination of OSI-906 and everolimus
  OSI-906: 100 mg Twice a Day, cycle-28 days
  Everolimus: 5mg Daily, cycle-28 days
  Interventions: Drug: OSI-906; Drug: Everolimus

INTERVENTIONS:
Drug: OSI-906 — Dose Level 1: 50 mg Twice a Day, cycle-28 days Dose Level 2: 100 mg Twice a Day, cycle-28 days Dose Level 2a: 100 mg Twice a Day, cycle-28 days
Drug: Everolimus — Dose Level 1: 5mg Daily, cycle-28 days Dose Level 2: 10mg Daily, cycle-28 days Dose Level 2a: 5mg Daily, cycle-28 days

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of the combination of OSI-906 and everolimus for the treatment of patients with refractory metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic cancer of the colon or rectum that has progressed on or for which the patient is intolerant to or not a candidate for: fluoropyrimidines, oxaliplatin, irinotecan, bevacizumab, and cetuximab or panitumumab.
* Testing for Kras mutation performed;Patients with mutated or wild type Kras are eligible.
* ECOG PS of 0-1
* Life expectancy of ≥ 3 months
* Adequate hematological function with ANC 1500, Platelets of 100,000, and hemoglobin of 9.0
* AST, ALT and Alk. Phos. ≤2.5 x ULN or ≤5 x ULN if known hepatic metastases and a total bilirubin ≤1.5 ULN
* Serum creatinine of ≤1.5 x ULN
* Fasting blood glucose <150 mg/dL
* Measurable disease according to RECIST 1.1
* Able to swallow whole pills
* INR ≤1.5 - Anticoagulation is allowed with LMW heparin
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤2.5 x ULN;If these thresholds are exceeded, the patient can be included after initiation of lipid lowering medication

Exclusion Criteria:

* Patients who have received any cancer therapies <4 weeks or 5 half lives (whichever is shorter) of initiating study therapy
* Treatment with any investigational drug ≤ 4 weeks, or 5 half-lives of the drug, whichever is shorter
* Patients who require coumadin for anticoagulation
* Patients who have had major surgery or significant traumatic injury ≤4 weeks of the of study treatment
* Minor surgery (with the exception of port placement) must be completed ≤ 7days prior to study therapy
* Previous treatment with an IGFR inhibitor or MTOR Inhibitor
* Chronic, systemic treatment with corticosteroids or another immunosuppressive agent
* Patients with QTc interval >450ms
* Patients who require drugs that can prolong QTc.
* Patients with congenital long QT syndrome, history of ventricular tachycardia, or ventricular fibrillation, or Torsades de Pointes with bradycardia.
* Immunization with attenuated live vaccines within 1 week of beginning study therapy or during study period;Close contact to anyone that has received live virus vaccine should be avoided
* Meningeal or brain metastasis
* Other malignancies < 3 years, with the exception of adequately treated basal or squamous cell carcinomas of the skin, or carcinoma in situ of the cervix
* Patients with known HIV
* Patients with positive testing for hepatitis B or C
* Patients with risk factors for hepatitis must be tested for hepatitis viral loadHepatitis risk factors include the following:

Lived in Asia, Africa, Central and South America, Eastern Europe, Spain, Portugal, and Greece Any blood transfusions before 1990 Any IV drug use Any dialysis Household contact with a Hep B infected patient Mother had Hep B High-risk sexual activity Body piercing/tattoos

* History suggestive of hepatitis B
* Any severe or uncontrolled conditions that could affect their study participation such as:Severely impaired lung function;DCLO ≤ 50% of normal predicted value;O² Sat <88% at rest on room air
* Congestive Heart Failure of NYHA Class III or IV
* Unstable angina, symptomatic CHF, MI ≤ 6 months, serious uncontrolled cardiac arrhythmia or any other clinically significant heart disease
* CVA, TIA, angioplasty, or cardiac stenting <12 months
* Ventricular arrhythmia requiring medication
* Known history of diabetes and/or patients who require ongoing use of insulin or oral anti-hyperglycemic therapy
* Known liver disease
* Impairment of GI function or gastrointestinal disease that in may significantly alter the absorption of study drugs
* Concurrent treatment with drugs that are strong CYP3A4 inducers or moderate/strong CYP3A4 inhibitors
* Concurrent treatment with drugs that are strong CYP1A2 inhibitors or inducers Women who are pregnant or breastfeeding.
* Concurrent severe, intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Bendell, MD, Study Chair — SCRI Development Innovations, LLC
Locations (2):
- United States (2):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Tennessee Oncology, Nashville, Tennessee

REFERENCES:
- [Derived] Bendell JC, Jones SF, Hart L, Spigel DR, Lane CM, Earwood C, Infante JR, Barton J, Burris HA. A phase Ib study of linsitinib (OSI-906), a dual inhibitor of IGF-1R and IR tyrosine kinase, in combination with everolimus as treatment for patients with refractory metastatic colorectal cancer. Invest New Drugs. 2015 Feb;33(1):187-93. doi: 10.1007/s10637-014-0177-3. Epub 2014 Oct 22. PMID 25335932

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 2a
Started | 7 | 6 | 5
Completed | 0 (Patients continued treatment until disease progression or unacceptable toxicity occurred.) | 0 (Patients continued treatment until disease progression or unacceptable toxicity occurred.) | 0 (Patients continued treatment until disease progression or unacceptable toxicity occurred.)
Not Completed | 7 | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 2a | Total
Number analyzed (Participants) | 7 | 6 | 5 | 18
Age, Continuous [Median (Full Range); unit: years] | 55 [47 to 73] | 54 [51 to 76] | 70 [44 to 76] | 55 [44 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 1 | 9
  Male | 3 | 2 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Maximum Tolerated Dose (MTD) of the Combination of OSI-906 and Everolimus for the Treatment of Patients With Refractory Metastatic Colorectal Cancer.
Description: The MTD of the drug combination will be determined as the highest dose at which ≤1 of 6 subjects experiences a Grade 3 or Grade 4 DLT according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0
Time Frame: 18 Months
Measure: Number; unit: milligrams
Groups:
- All Patients: Determination of the MTD consists of the selection of one of the three dose levels as the maximum tolerated dose. This outcome is the same for all patients.
Arm/Group | All Patients
Number analyzed (Participants) | 18
milligrams
  OSI-906 BID Dose | 50
  Everolimus QD Dose | 5

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time between Day 1 Cycle 1 and date of first documented recurrence or death. Patients who do not exhibit progression while on trial will be censored at their last known assessment. Progression is defined per RECIST criteria as either 1) at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest (nadir) sum since the treatment started, or the appearance of one or more new lesions. Requires not only 20% increase, but absolute increase of a minimum of 5 mm over sum. OR 2) Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: 18 Months
Measure: Mean (Standard Deviation); unit: months
Groups:
- Dose Level 1: combination of OSI-906 (50 mg Twice a Day, cycle-28 days) and everolimus (5mg Daily, cycle-28 days)
- Dose Level 2: combination of OSI-906 (100 mg Twice a Day, cycle-28 days) and everolimus (10 mg Daily, cycle-28 days)
- Dose Level 2a: combination of OSI-906 (100 mg Twice a Day, cycle-28 days) and everolimus (5 mg Daily, cycle-28 days)
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 2a
Number analyzed (Participants) | 7 | 6 | 5
months | 2.8 (1) | 3.6 (5.2) | 1.6 (0.5)

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time between Day 1 Cycle 1 to the date of death from any cause. Those remaining alive will be censored at their last known assessment or follow-up.
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: weeks
Groups:
- Dose Level 1: combination of OSI-906 (50 mg Twice a Day, cycle-28 days) and everolimus (5 mg Daily, cycle-28 days)
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 2a
Number analyzed (Participants) | 7 | 6 | 5
weeks | 5.1 (2.4) | 5.1 (5) | 3.3 (2.4)

4. Secondary Outcome: Response Rate
Description: Response rate (RR) will be estimated as the proportion of patients exhibiting complete response or partial response out of all evaluable cases. Complete Response is defined per RECIST as disappearance of all target/non-target lesions and normalization of tumor markers. Partial Response is defined per RECIST as At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: 18 months
Population: Only patients who received at least 8 weeks of treatment were considered evaluable for response and were included in the response rate analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 2a
Number analyzed (Participants) | 6 | 1 | 3
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 18 months
Description: All patients who received at least one dose of protocol treatment were followed for safety. Adverse events and serious adverse events were collected from the day of the first dose to 30 days after the last dose of the study medication and graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Groups:
- Dose Level 2a: combination of OSI-906 (50 mg Twice a Day, cycle-28 days) and everolimus (5 mg Daily, cycle-28 days)
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 2a
Serious Adverse Events (participants affected / at risk) | 2/7 | 1/6 | 2/5
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=7) | Dose Level 2 (N=6) | Dose Level 2a (N=5)
Gastrointestinal disorders - Other, esophageal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, mechanical bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, disease progression (General disorders) | 0 | 1 (1) | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia with Bleeding (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=7) | Dose Level 2 (N=6) | Dose Level 2a (N=5)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (7) | 2 (3) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis (Gastrointestinal disorders) | 0 (0) | 3 (7) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (3) | 3 (3) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (2) | 3 (3) | 0 (0)
Frequent stools (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Green/dark brown stools (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (9) | 2 (4) | 2 (3)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Difficulty sleeping (General disorders) | 1 (1) | 0 (0) | 0 (0)
Edema: head and neck (General disorders) | 1 (1) | 0 (0) | 0 (0)
Edema: limb (General disorders) | 1 (1) | 0 (0) | 0 (0)
facial stuffiness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage (General disorders) | 0 (0) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Elevated bilirubin (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 1 (1) | 0 (0)
ALT elevated (Investigations) | 1 (1) | 0 (0) | 0 (0)
AST elevated (Investigations) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC (GU) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 4 (6) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased urine output (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Clear/blood tinged drainage (sinus congestion) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Coughing up blood (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (2) | 1 (1)
Cold sore (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
generalized itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Laceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth soreness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dry/swollen sinus (General disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Neutrophils decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Pain - Chest tightness (General disorders) | 1 (2) | 0 (0) | 0 (0)
Pain - Lower back (General disorders) | 1 (3) | 0 (0) | 0 (0)
Pain - lumbar back (General disorders) | 0 (0) | 1 (2) | 0 (0)
Pain (anal) (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (gastrointestinal) (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (GU) (General disorders) | 0 (0) | 1 (1) | 0 (0)
pain (musculoskeletal) (General disorders) | 1 (1) | 2 (2) | 0 (0)
Pain (neurology) (General disorders) | 0 (0) | 1 (1) | 0 (0)
Runny nose (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (General disorders) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Investigations) | 0 (0) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites